CLINICAL TRIAL: NCT01536015
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Effect of Rotigotine on Motor Symptoms in Patients With Advanced Parkinson's Disease With Motor Fluctuations and Symptoms of Gastrointestinal Dysfunction
Brief Title: Effect of Rotigotine on Motor Symptoms in Patients With Advanced Parkinson's Disease (PD) With Motor Fluctuations and Symptoms of Gastrointestinal Dysfunction
Acronym: ROADMAP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped due to low enrollment.
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP1055
Record Dates: First submitted 2012-02-15; First posted 2012-02-20 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Advanced Parkinson's Disease
Keywords: Rotigotine; Neupro®; Levodopa; Gastrointestinal Dysfunction
MeSH Terms: interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine (Experimental): Rotigotine patch titrated from 4 mg/24 h - 8 mg/24 h or until effective or maximum dose is reached.
  Interventions: Drug: Rotigotine
- Placebo (Placebo Comparator): Placebo patch.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rotigotine — Strength and Form: 4 - 8 mg patches, one patch applied every 24 hours
  Dosage and Frequency: One patch every 24 hours
  Duration: 10 weeks
  Other Names: Neupro®
  Arms: Rotigotine
Drug: Placebo — Frequency: One patch applied every 24 hours
  Duration: 10 weeks
  Arms: Placebo

SUMMARY:
The primary purpose is to demonstrate superiority of Rotigotine over Placebo on motor symptoms when used in subjects with symptoms of Gastrointestinal Dysfunction. Hypothesis: Rotigotine will decrease OFF time compared to Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject is informed and given ample time and opportunity to think about his/her participation in this study and has given his/her written informed consent on an Institutional Review Board approved consent form
* Subject is willing and able to comply with all study requirements (protocol, visit schedule, procedures, and medication application)
* Subject is male or female and ≥ 30 years of age
* Subject has Idiopathic Parkinson's Disease of more than 3 years duration, as defined by the cardinal sign, bradykinesia, plus the presence of at least 1 of the following: resting tremor, rigidity, impairment of postural reflexes; and is without any other known or suspected cause of Parkinsonism
* Subject has a Hoehn & Yahr stage score II through IV
* Subject must be on a stable dose of L-dopa, either short-acting or sustained release (in combination with Benserazide or Carbidopa), of at least 200 mg/day administered in at least 2 intakes, for at least 21 days prior to starting Parkinson's diaries
* Subject must be able to differentiate between the "on" and "off" state (and thereby be able to recognize the Time To "On" (TTON)), and be willing and able to accurately complete a Parkinson's Disease subject diary on designated days (with assistance from caregivers, if required)
* Subject must complete 6 Parkinson's diaries over a period of 6 days, with 4 of the 6 Parkinson's diaries being "valid" as determined by the investigator. The "valid" Parkinson's diaries confirm that the subject has an average of at least 2.5 h/day spent in the "off" state
* Subject receiving a Monoamine Oxidase (MAO)-B Inhibitor (eg, Selegiline or Rasagiline), an n-Methyl-d-Aspartate Antagonist (eg, Amantadine), or allowed anti-Parkinson medications and has been on a stable dose for at least 21 days prior to starting Parkinson's diaries and is anticipated to be maintained on that dose for the duration of the study
* Subject has clinical symptoms of Gastrointestinal Dysfunction (GID) confirmed by at least 1 of the following

  •Parkinson's disease-related GI symptoms as per the Gastrointestinal Degenerative Scale (GIND) Scale: defecatory dysfunction, constipation, excessive gas, abdominal pain, bloating, nausea, vomiting, anorexia, early satiety, or weight loss (except sialorrhea and dysphagia)
* Female subjects of childbearing potential must agree to use 1 of the following contraceptive methods: oral contraceptive, intrauterine device, or double-barrier method, throughout the study and for 2 weeks after the removal of study medication

Exclusion Criteria:

* Subject has previously participated in this study
* Subject has participated in another study of an investigational medicinal product (IMP) or a medical device within the last 30 days or is currently participating in another study of an IMP or a medical device
* Subject has an Atypical Parkinsonian Syndrome due to drugs (eg, Metoclopramide, Flunarizine), Metabolic Neurogenetic Disorders (eg, Wilson's Disease), Encephalitis, Cerebrovascular Disease, or Degenerative Disease (eg, Progressive Supranuclear Palsy)
* Subject has a history of Pallidotomy, Thalamotomy, Deep Brain Stimulation, or Fetal Tissue Transplant
* Subject has Dementia, Active Psychosis, or Hallucinations
* Subject exhibits Dopaminergic Dysregulation Syndrome
* Subject is receiving therapy with certain medications in a specific timeframe as specified in the protocol
* Subject has history of chronic Gastrointestinal (GI) Disease not related to Parkinson's disease which in the judgement of the investigator may affect the ability of the subject to participate in the study (ie, Irritable Bowel Syndrome, Diverticulitis, Crohn's Disease, etc) or GI/abdominal surgery (except for Appendectomy, Hysterectomy, or Cholecystectomy)
* Subject has had any GI surgery in the 3 months prior to the Screening Visit
* Subject has a current diagnosis of Epilepsy, has a history of seizures as an adult, or has a history of stroke or Transient Ischemic Attack within 1 year prior to the Screening Visit
* Subject has clinically relevant Hepatic or Renal Dysfunction
* Subject has clinically relevant Cardiac Dysfunction (any cardiac disorder that in the opinion of the investigator would put the subject at risk of clinically relevant arrhythmia)
* Subject has had a Myocardial Infarction within the last 1 year prior to the Screening Visit
* Subject has a history of Symptomatic (not Asymptomatic) Orthostatic Hypotension
* Subject has a Systolic Blood Pressure (BP) < 105 mmHg at the Screening Visit
* Subject has a history of chronic alcohol or drug abuse within the prior 6 months
* Female subject is pregnant or lactating
* Subject (male or female) is of child bearing potential but not surgically sterile or not using adequate birth control methods
* Subject has evidence of an Impulse Control Disorder according to the Modified Minnesota Impulsive Disorders Interview (mMIDI) at the Screening Visit
* Subject has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ('Yes') to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at the Screening Visit
* Subject has a significant skin disease/condition that would make transdermal drug use inappropriate, including a history of skin sensitivity to adhesives or other transdermal medications
* Subject has a known hypersensitivity to any components of the Rotigotine patch, including Sodium Metabisulfite
* Subject has any medical, psychiatric, or cognitive condition, or laboratory abnormality that would, in the opinion of the investigator, jeopardize or compromise the subject's well-being or ability to participate in the study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — 877-822-9493
Locations (26):
- United States (26):
  - 011, Birmingham, Alabama
  - 001, Gilbert, Arizona
  - 022, Fountain Valley, California
  - 017, Irvine, California
  - 028, Pasadena, California
  - 015, Sunnyvale, California
  - 008, Gainesville, Florida
  - 009, Miami, Florida
  - 010, Ormond Beach, Florida
  - 006, Sunrise, Florida
  - 032, Annapolis, Maryland
  - 027, Lincoln, Nebraska
  - 016, Commack, New York
  - 026, Mineola, New York
  - 034, Charlotte, North Carolina
  - 002, Raleigh, North Carolina
  - 007, Salisbury, North Carolina
  - 021, Toledo, Ohio
  - 023, Tulsa, Oklahoma
  - 031, Cordova, Tennessee
  - 018, Memphis, Tennessee
  - 014, Houston, Texas
  - 030, Richmond, Virginia
  - 003, Virginia Beach, Virginia
  - 012, Kirkland, Washington
  - 013, Milwaukee, Wisconsin

REFERENCES:
- See also: FDA safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The total duration of the study was to be a maximum of 19 weeks for each subject, including the Screening Period (within 50 days prior to Day 1), the Titration Period (up to 3 weeks), the Maintenance Period (up to 7 weeks), and a Safety Follow-Up Visit. The Participant Flow refers to the Randomized Set which includes all randomized subjects.
Pre-assignment Details: A total of approximately 150 subjects were planned to be randomized in a 1:1 ratio to either Rotigotine or Placebo.
Groups:
- Placebo: Placebo patch
  Placebo: Frequency: One patch applied every 24 hours
  Duration: 10 weeks
- Rotigotine: Rotigotine patch titrated from 4 mg/24 h - 8 mg/24 h or until effective or maximum dose is reached.
  Rotigotine: Strength and Form: 4 - 8 mg patches, one patch applied every 24 hours
  Dosage and Frequency: One patch every 24 hours
  Duration: 10 weeks
Period: Overall Study
Arm/Group | Placebo | Rotigotine
Started | 12 | 13
Completed | 4 | 3
Not Completed | 8 | 10
Not completed — Adverse Event | 1 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Inclusion Criterion not met | 2 | 0
Not completed — Study closure | 5 | 5

BASELINE CHARACTERISTICS:
Population: The Analysis Population Description refers to the Safety Set (SS) which consists of all randomized subjects who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rotigotine | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (8.2) [52 to 78] | 66.7 (9.6) [51 to 82] | 66.4 (8.8) [51 to 82]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 7 | 7 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 11 | 8 | 19
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25
Weight [Mean (Standard Deviation); unit: kilogram] | 84.64 (14.93) [65.8 to 112.4] | 76.67 (19.53) [49.4 to 121.6] | 80.50 (17.58) [49.4 to 121.6]
Height [Mean (Standard Deviation); unit: centimeter] | 171.79 (13.65) [149.9 to 198.4] | 173.86 (10.61) [157.5 to 192.0] | 172.87 (11.95) [149.9 to 198.4]
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram/m^2] | 28.714 (4.167) [21.48 to 37.30] | 25.113 (4.809) [19.81 to 35.36] | 26.842 (4.785) [19.81 to 37.30]

OUTCOME MEASURES:

1. Primary Outcome: Change in Rotigotine Versus Placebo in the Absolute Time Spent "Off" From Baseline to the End of the 7-week Maintenance Period
Description: Mean number of hours marked "off" during a 24-hour period.
Time Frame: Baseline to 10 weeks
Population: This study was terminated early because of low enrollment. Due to the early termination no analysis tables of efficacy data were done and no descriptive summaries of efficacy data were produced.
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS UPDRS) Part III (Motor Examination) in the "on" State From Baseline to the End of the 7-week Maintenance Period
Description: The Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS UPDRS) Part III is an 18-item scale with each single item of the scale ranging from 0 (normal) to 4 (severe).
Time Frame: Baseline to 10 weeks
Population: as for outcome 1
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Predictability of "Off" Time (Using MDS UPDRS Part IV Item 4.5) From Baseline to End of the 7-week Maintenance Period
Description: The Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS UPDRS) Part IV is a 6-item scale with each single item of the scale ranging from 0 (normal) to 4 (severe).
Time Frame: Baseline to 10 weeks
Population: as for outcome 1
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Score on Gastrointestinal Neurodegenerative Scale (GIND) From Baseline to the End of the of the 7-week Maintenance Period
Description: Gastrointestinal Neurodegenerative Scale (GIND) is an 18-item scale measuring gastrointestinal dysfunction with each single item of the scale ranging from 0 (never or not at all) to 5 (very severe).
Time Frame: Baseline to 10 weeks
Population: as for outcome 1
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Score on Fatigue Severity Scale (FSS) From Baseline to the End of 7-week Maintenance Period
Description: The Fatigue Severity Scale is a 9-item scale measuring the impact of fatigue on everyday functioning (e.g. "fatigue interferes with my work, each single item of the scale ranging from 1 (disagree) to 7 (agree).
Time Frame: Baseline to 10 weeks
Population: as for outcome 1
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Score on Parkinson's Disease Questionnaire (PDQ8) From Baseline to the End of 7-week Maintenance Period
Description: The Parkinson's Disease Questionnaire (PDQ-8) is a self-administered 8-item questionnaire that assesses issues associated with Parkinson's disease. Each single item of the 8-item questionnaire ranges from 0 (never) to 4 (always).
Time Frame: Baseline to 10 weeks
Population: as for outcome 1
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From Screening (Day -50 to Day -1) up to the Safety Follow-up Visit (14±2 days after the End of Maintenance/Start of De-Escalation Visit or Premature Withdrawal/Start of De-Escalation Visit).
Description: Only Treatment Emergent Adverse Events were reported. The Analysis Population refers to the Safety Set (SS). The SS consists of all randomized subjects who received at least 1 dose of study medication.
Arm/Group | Placebo | Rotigotine
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/13
Other Adverse Events (participants affected / at risk) | 4/12 | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Rotigotine (N=13)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Rotigotine (N=13)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
Dyskinesia (Nervous system disorders) | 1 (1) | 2 (5)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days